CLINICAL TRIAL: NCT04773665
Title: A Phase 1a/1b, Randomized, Observer-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of the COVID-19 (SARS-CoV-2) Vaccine Candidates VBI-2902a and VBI-2905a in Healthy Adults
Brief Title: Safety, Tolerability, and Immunogenicity of the COVID-19 Vaccine Candidates VBI-2902a and VBI-2905a
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VBI Vaccines Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: VBI-2902a-CT01
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Covid19
Keywords: enveloped virus-like particle (eVLP); SARS-CoV-2 spike; neutralizing antibody; cell-mediated immune responses
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is an observer-blinded study. Both participants and the study center staff performing outcome measurement are blinded; vaccines will be administered by qualified unblinded study personnel who have no other role in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase 1a, Group G1 (Experimental): 20 participants age 18-54 will receive VBI-2902a at a dose of 5 μg of S protein at Day 1 and placebo at Day 28
  Interventions: Biological: VBI-2902a; Biological: Placebo
- Phase 1a, Group G2 (Experimental): 20 participants age 18-54 will receive VBI-2902a at a dose of 5 μg of S protein at Days 1 and 28
  Interventions: Biological: VBI-2902a
- Phase 1a, Group G3 (Placebo Comparator): 20 participants age 18-54 will receive placebo at Days 1 and 28
  Interventions: Biological: Placebo
- Phase 1b, Group G4 (Experimental): 27 participants age 18-54 will receive VBI-2905a at a dose of 5 μg of S protein at Day 1
  Interventions: Biological: VBI-2905a
- Phase 1b, Group G5 (Placebo Comparator): 27 participants age 18-54 will receive placebo at Day 1
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VBI-2902a — VBI-2902a is an intramuscular injection of VBI-2902a investigational enveloped virus-like particle COVID-19 vaccine with aluminum phosphate adjuvant.
  Arms: Phase 1a, Group G1; Phase 1a, Group G2
Biological: Placebo — 0.9% sodium chloride
  Arms: Phase 1a, Group G1; Phase 1a, Group G3; Phase 1b, Group G5
Biological: VBI-2905a — VBI-2905a is an intramuscular injection of VBI-2905a investigational enveloped virus-like particle COVID-19 vaccine with aluminum phosphate adjuvant.
  Arms: Phase 1b, Group G4

SUMMARY:
VBI-2902a and VBI-2905a are investigational vaccine candidates that use enveloped virus-like particle (eVLP) expression of a modified version of the SARS-CoV-2 spike (S) glycoprotein and are designed to induce neutralizing antibody and cell-mediated immune responses against the SARS-CoV-2 spike protein. VBI-2902a expresses the spike protein of SARS-CoV-2 Wuhan isolate (the first virus variant isolated in 2019 in Wuhan, China), while VBI-2905a expresses the spike protein of SARS-CoV-2 variant Beta (B.1.351 variant, first isolated in 2020 in South Africa).

The Phase 1a portion of this study tests one- and two-dose regimens of VBI- 2902a with 5 μg S protein content and aluminum phosphate (alum) adjuvant or placebo delivered by intramuscular (IM) injection. The Phase 1b portion of the study tests a one-dose regimen of VBI-2905a with 5 μg S protein content and alum adjuvant or placebo delivered by IM injection in participants previously vaccinated with an authorized mRNA COVID-19 vaccine.

DETAILED DESCRIPTION:
Phase 1a:

The primary objective is to evaluate the safety and tolerability of VBI-2902a containing 5 μg of S protein in one- or two-dose regimens in healthy adults of 18-54 years of age.

The secondary objective is to evaluate the immunogenicity of VBI-2902a containing 5 μg of S protein in one- or two-dose regimens in healthy adults 18-54 years of age.

* Group G1 - 20 participants will receive VBI-2902a at a dose of 5 μg of S protein at Day 1 and placebo at Day 28.
* Group G2 - 20 participants will receive VBI-2902a at a dose of 5 μg of S protein at Days 1 and 28.
* Group G3 - 20 participants will receive placebo at Days 1 and 28.

An Independent Data Safety Monitoring Board (DSMB) will review blinded safety data (reactogenicity, adverse events (AEs) and safety laboratory assessments) at Day 7 after the first vaccination. The second vaccination will only be given if the DSMB confirms that Day 7 safety is acceptable and that stopping rules were not met. The DSMB will further review blinded post-vaccination safety through Day 35, 7 days after the second vaccination and through Day 56, 28 days after the second vaccination. The study will be unblinded following DSMB review of safety data collected through Day 56. Study participants will continue with study visits as planned up to 12 months of follow up after the first dose of study vaccine.

Phase 1b:

The primary objective is to evaluate the safety and tolerability of a one-dose regimen of VBI-2905a at a 5 μg dose level of S protein in healthy adults (age 18-54 years) who had been previously vaccinated with mRNA vaccines.

The secondary objective is to evaluate the immunogenicity of a one-dose regimen of VBI-2905a at a 5 μg dose level of S protein in healthy adults (age 18-54 years) who had been previously vaccinated with mRNA vaccines.

A total of 54 healthy adults, age 18-54 years, with no history of clinical or laboratory diagnosis of SARS-CoV- 2 infection or COVID-19 illness, will be enrolled in the Phase 1b part of the study. All participants in Phase 1b will have been previously vaccinated with an authorized mRNA COVID-19 vaccine, including the second dose administered at least 4 months prior to enrollment, will be randomized at a 1:1 ratio to receive, in a blinded fashion, one dose of VBI-2905a or placebo:

* Group G4 - 27 participants will receive VBI-2905a at a dose of 5 μg of S protein at Day 1
* Group G5 - 27 participants will receive placebo at Day 1

The DSMB will review blinded post-vaccination safety data 7 days after each vaccination (reactogenicity, AEs and safety laboratory assessments). In Phase 1b, the DSMB will review blinded Day 7 safety data after the first 10 participants in groups G4 and G5 have received the first dose. Only after the DSMB confirms that safety is acceptable and that stopping rules were not met will the enrollment in the respective study groups continue to its completion.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, each participant must satisfy all of the following criteria:

1. Healthy female and male participants 18 -54 years of age.
2. If female:

   1. is of childbearing potential and must have a negative pregnancy test prior to study vaccinations and agree to use an effective method of birth control as deemed appropriate by the investigator (e.g., hormonal contraceptive, barrier contraceptive with additional spermicide, or an intrauterine device) beginning >30 days prior to the first study vaccine administration and continuing until the end of the study.

      OR
   2. is not of childbearing potential, defined as postmenopausal (12 months with no menses without an alternative medical cause) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy orhysterectomy).
3. Phase 1b: previously received a full course (2 doses) of an authorized S protein mRNA COVID-19 vaccine (e.g. COVID-19 vaccines produced by Pfizer/BioNTech or Moderna) at least 4 months prior to enrollment.
4. Sign an informed consent document indicating understanding of the purpose of and procedures required for the study and willingness to participate in the study.

Exclusion Criteria

Participants with any of the following criteria will be excluded:

1. History of clinical or laboratory diagnosis of COVID-19 or SARS-CoV-2 infection.
2. Phase 1b: Previous receipt of an experimental or authorized SARS-CoV-2 (COVID-19) vaccines other than an S-protein mRNA vaccine.
3. Phase 1a: Previous receipt of an experimental or authorized SARS-CoV-2 (COVID-19) vaccine.
4. Positive PCR or rapid antigen test for SARS-CoV-2 at screening.
5. Individuals with chronic medical conditions, including any of the following:

   1. Diabetes mellitus Type 1 or Type 2
   2. Chronic pulmonary disease (e.g., COPD or Asthma)
   3. Hypertension (e.g., SBP >140 mmHg or DBP >90 mmHg)
   4. Chronic kidney disease (e.g., GFR <60 mL/min/1.73 m2)
   5. Chronic liver disease
   6. Obesity (e.g., BMI >30 kg/m2)
6. Any history of cancer requiring chemotherapy or radiation within 5years.
7. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
8. Lack of participant's capacity (mental, social, behavioral), in the investigator's judgement, to provide informed consent for participation in the study.
9. Known or suspected impairment of immunological function, including but not limited to autoimmune diseases:

   1. autoimmune diseases (e.g. multiple sclerosis, type 1 diabetes, myasthenia gravis, Crohn disease and other inflammatory bowel diseases, celiac disease, systemic lupus erythematosus, scleroderma, including diffuse systemic form and CREST syndrome, systemic sclerosis, dermatomyositis polymyositis, rheumatoid arthritis, juvenile idiopathic arthritis, autoimmune thyroiditis - including Hashimoto thyroiditis, Grave's or Basedow's disease, immune thrombocytopenic purpura, autoimmune hemolytic anemia, autoimmune hepatitis, psoriasis, vitiligo, vasculitis, Guillain- Barré syndrome, Transverse myelitis, Addison's disease, Bell's Palsy and Alopecia Areata);
   2. secondary immunodeficiency disorders (e.g., Acquired Immunodeficiency Syndrome caused by Human Immunodeficiency Virus infection (HIV/AIDS), solid organ transplant,splenectomy);
   3. primary immunodeficiency disorders (e.g., common variable immune deficiency (CVID), Defective phagocytic cell function and neutropenia syndromes, complement deficiency).
10. History of allergic reactions or anaphylactic reaction to any vaccine component.
11. Known infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
12. Pregnant or breastfeeding or plans to conceive from 2 weeks before the study until the end of study.
13. Clinically significant abnormal physical examination, vital signs, or clinically significant abnormal values for hematology, serum chemistry or urinalysis at screening as determined by the investigator.
14. Any laboratory test abnormality that would be considered of Grade 1 severity or above (as per FDA grading guidelines) and is considered as clinically significant by the investigator. Grade 2 severity or above is exclusionary, regardless of clinical assessment.
15. Has received blood products or immunoglobulin within 90 days of enrollment or is likely to require blood products during the study period.
16. Chronic administration (defined as more than 14 days in total) of immune-suppressive or other immune-modifying drug within six months prior to the product dose (for corticosteroids, this is defined as prednisone ≥20 mg/day or equivalent). Inhaled and topical steroids are allowed.
17. Immunization with attenuated vaccines (e.g., measles, mumps, and rubella vaccine) within 4 weeks prior to enrollment.
18. Immunization with inactivated vaccines (e.g., influenza) within 2 weeks prior to enrolment.
19. Participation in another clinical study within 30 days.
20. Any skin abnormality or tattoo that would limit post-vaccination injection site assessment.
21. Family members of study site personnel.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne M Langley, MD, Principal Investigator — Canadian Center for Vaccinology; William Cameron, MD, Principal Investigator — Ottawa Hospital
Locations (4):
- Canada (4):
  - Canadian Center for Vaccinology, Halifax, Nova Scotia
  - Ottawa Hospital, Ottawa, Ontario
  - LMC Manna - Bayview CPU, Toronto, Ontario
  - Manna Toronto, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1a, Group G1: Previously unvaccinated participants received VBI-2902a at a dose of 5 μg of S protein at Day 1 and placebo at Day 28
  VBI-2902a: VBI-2902a is an intramuscular injection of VBI-2902a investigational enveloped virus-like particle COVID-19 vaccine with aluminum phosphate adjuvant.
  Placebo: 0.9% sodium chloride
- Phase 1a, Group G2: Previously unvaccinated participants received VBI-2902a at a dose of 5 μg of S protein at Days 1 and 28
  VBI-2902a: VBI-2902a is an intramuscular injection of VBI-2902a investigational enveloped virus-like particle COVID-19 vaccine with aluminum phosphate adjuvant.
- Phase 1a, Group G3: Previously unvaccinated participants received placebo at Days 1 and 28
  Placebo: 0.9% sodium chloride
- Phase 1b, Group G4: Previously vaccinated participants received VBI-2905a at a dose of 5 μg of S protein at Day 1
  VBI-2905a: VBI-2905a is an intramuscular injection of VBI-2905a investigational enveloped virus-like particle COVID-19 vaccine with aluminum phosphate adjuvant.
- Phase 1b, Group G5: Previously vaccinated participants received placebo at Day 1
  Placebo: 0.9% sodium chloride
Period: Overall Study
Arm/Group | Phase 1a, Group G1 | Phase 1a, Group G2 | Phase 1a, Group G3 | Phase 1b, Group G4 | Phase 1b, Group G5
Started | 21 | 20 | 20 | 27 | 26
Completed | 19 | 19 | 19 | 24 | 26
Not Completed | 2 | 1 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1a, Group G1 | Phase 1a, Group G2 | Phase 1a, Group G3 | Phase 1b, Group G4 | Phase 1b, Group G5 | Total
Number analyzed (Participants) | 21 | 20 | 20 | 27 | 26 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (9.37) | 32.9 (9.45) | 30.8 (9.03) | 36.3 (11.03) | 36.6 (9.87) | 33.68 (9.77)
Age, Customized [Count of Participants; unit: Participants]
  18 to 39 | 17 | 15 | 18 | 14 | 15 | 79
  40 to 55 | 4 | 5 | 2 | 13 | 11 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 11 | 16 | 16 | 57
  Male | 14 | 13 | 9 | 11 | 10 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2 | 2 | 2 | 1 | 2 | 9
  Race: Black or African American | 0 | 0 | 2 | 0 | 0 | 2
  Race: First Nations | 0 | 0 | 0 | 0 | 0 | 0
  Race: Multiple | 1 | 0 | 1 | 1 | 3 | 6
  Race: White | 16 | 17 | 12 | 24 | 21 | 90
  Race: Other | 2 | 1 | 3 | 1 | 0 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 1 | 1 | 1 | 1 | 0 | 4
  Ethnicity: Not Hispanic or Latino | 20 | 19 | 19 | 26 | 26 | 110
Region of Enrollment [Number; unit: participants]
  Canada | 21 | 20 | 20 | 27 | 26 | 114

OUTCOME MEASURES:

1. Primary Outcome: Rate of Local Solicited Adverse Events After Each Study Vaccination
Description: The occurrence of local (near injection site) adverse events actively solicited from the participant during the post-administration follow-up period.
  An adverse event is defined as any untoward medical occurrence in a participant administered a pharmaceutical product. It does not necessarily have to have a causal relationship with this treatment. An adverse event can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product whether or not considered related to the medicinal product.
Time Frame: Through 7 days after each study vaccination
Population: Safety Set: subjects who received a study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a, Group G1 | Phase 1a, Group G2 | Phase 1a, Group G3 | Phase 1b, Group G4 | Phase 1b, Group G5
Number analyzed (Participants) | 21 | 20 | 20 | 27 | 26
Participants
  Any local solicited adverse event | 13 | 17 | 11 | 23 | 8
  Pain | 11 | 17 | 10 | 20 | 4
  Tenderness | 10 | 13 | 9 | 19 | 6
  Itchiness | 2 | 0 | 2 | 2 | 1
  Erythema/redness | 0 | 0 | 0 | 0 | 1
  Induration/swelling | 0 | 1 | 0 | 1 | 0

2. Primary Outcome: Rate of Systemic Solicited Adverse Events After Each Study Vaccination
Description: The occurrence of systemic adverse events actively solicited from the participant during the post-administration follow-up period.
  An adverse event is defined as any untoward medical occurrence in a participant administered a pharmaceutical product. It does not necessarily have to have a causal relationship with this treatment. An adverse event can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product whether or not considered related to the medicinal product.
Time Frame: Through 7 days after each study vaccination
Population: Safety Set: subjects who received a study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a, Group G1 | Phase 1a, Group G2 | Phase 1a, Group G3 | Phase 1b, Group G4 | Phase 1b, Group G5
Number analyzed (Participants) | 21 | 20 | 20 | 27 | 26
Participants
  Any systemic solicited adverse event | 15 | 15 | 15 | 15 | 16
  Fatigue | 12 | 12 | 10 | 10 | 8
  Diarrhoea | 5 | 1 | 4 | 1 | 4
  Nausea/vomiting | 1 | 1 | 3 | 2 | 3
  Headache | 9 | 10 | 8 | 7 | 10
  Myalgia | 8 | 6 | 6 | 4 | 4
  Fever | 0 | 0 | 2 | 0 | 0

3. Primary Outcome: Rate of Unsolicited Adverse Events After Each Study Vaccination
Description: Any adverse event reported in addition to those solicited during the clinical study.
  An adverse event is defined as any untoward medical occurrence in a participant administered a pharmaceutical product. It does not necessarily have to have a causal relationship with this treatment. An adverse event can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product whether or not considered related to the medicinal product.
Time Frame: Through 28 days after each study vaccination
Population: Safety Set: subjects who received a study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a, Group G1 | Phase 1a, Group G2 | Phase 1a, Group G3 | Phase 1b, Group G4 | Phase 1b, Group G5
Number analyzed (Participants) | 21 | 20 | 20 | 27 | 26
Participants
  Any unsolicited AE | 11 | 12 | 10 | 7 | 7
  Palpitations | 1 | 0 | 0 | 1 | 0
  Eye pruritus | 0 | 1 | 0 | 0 | 0
  Dyspepsia | 0 | 1 | 0 | 0 | 0
  Nausea | 1 | 0 | 0 | 0 | 0
  Paraesthesia oral | 0 | 0 | 1 | 0 | 0
  Chest pain | 1 | 0 | 0 | 0 | 0
  Chills | 1 | 0 | 1 | 0 | 0
  Fatigue | 2 | 1 | 3 | 0 | 0
  Injection site bruising | 1 | 2 | 0 | 0 | 0
  Injection site haemorrhage | 0 | 0 | 1 | 0 | 0
  Injection site pain | 0 | 1 | 0 | 0 | 0
  Pain | 1 | 0 | 0 | 0 | 0
  Pyrexia | 1 | 0 | 1 | 0 | 0
  Vaccination site pain | 3 | 0 | 1 | 0 | 4
  Vaccination site reaction | 0 | 1 | 1 | 0 | 0
  COVID-19 | 2 | 0 | 1 | 0 | 0
  Oral herpes | 1 | 0 | 1 | 0 | 0
  Pharyngitis | 1 | 0 | 0 | 0 | 0
  Rhinitis | 1 | 0 | 0 | 0 | 0
  Urinary tract infection | 0 | 1 | 1 | 0 | 0
  Arthropod bite | 0 | 2 | 0 | 0 | 0
  Limb injury | 0 | 1 | 0 | 0 | 0
  Aspartate aminotransferase increased | 1 | 0 | 0 | 0 | 0
  Blood bilirubin increased | 0 | 0 | 1 | 0 | 0
  Gamma-glutamyltransferase decreased | 0 | 0 | 1 | 0 | 0
  Liver function test increased | 0 | 0 | 1 | 0 | 0
  Lymph node palpable | 0 | 0 | 1 | 0 | 0
  Arthralgia | 1 | 0 | 2 | 0 | 0
  Joint stiffness | 1 | 0 | 0 | 0 | 0
  Muscular weakness | 0 | 0 | 1 | 0 | 1
  Myalgia | 1 | 1 | 0 | 0 | 0
  Dizziness | 0 | 1 | 0 | 0 | 0
  Headache | 2 | 1 | 2 | 1 | 1
  Anxiety | 1 | 0 | 0 | 0 | 0
  Vaginal haemorrhage | 0 | 1 | 0 | 0 | 0
  Cough | 0 | 0 | 1 | 1 | 0
  Dyspnoea | 0 | 1 | 0 | 0 | 0
  Nasal congestion | 2 | 0 | 1 | 0 | 0
  Rhinorrhoea | 0 | 0 | 1 | 0 | 1
  Throat tightness | 0 | 1 | 0 | 0 | 0
  Alopecia | 0 | 1 | 0 | 0 | 0
  Eustachian tube obstruction | 0 | 0 | 0 | 1 | 0
  Tinnitus | 0 | 0 | 0 | 1 | 0
  Vertigo | 0 | 0 | 0 | 1 | 0
  Abdominal pain | 0 | 0 | 0 | 1 | 0
  Flatulence | 0 | 0 | 0 | 1 | 0
  Alcohol poisoning | 0 | 0 | 0 | 1 | 0
  Haemoglobin decreased | 0 | 0 | 0 | 1 | 0
  Neutrophil count decreased | 0 | 0 | 0 | 1 | 0
  White blood cell count decreased | 0 | 0 | 0 | 1 | 0
  Bone pain | 0 | 0 | 0 | 1 | 0
  Muscle fatigue | 0 | 0 | 0 | 0 | 1
  Musculoskeletal stiffness | 0 | 0 | 0 | 1 | 0
  Neck pain | 0 | 0 | 0 | 0 | 1
  Pain in extremity | 0 | 0 | 0 | 1 | 0
  Heavy menstrual bleeding | 0 | 0 | 0 | 1 | 0
  Menstruation irregular | 0 | 0 | 0 | 1 | 0
  Oligomenorrhoea | 0 | 0 | 0 | 1 | 0
  Oropharyngeal pain | 0 | 0 | 0 | 0 | 1

4. Secondary Outcome: Geometric Mean Titer (GMT) of Neutralizing Antibody in Serum (Phase 1a)
Description: Virus-neutralizing antibody titers in serum were determined at baseline and post-vaccination using a pseudovirus neutralization assay (PNA). Titers are expressed as the highest serum dilution neutralizing 50% of viral infectivity (PNA50). Neutralization was tested against pseudoviruses expressing the spike protein of the ancestral (Wuhan) SARS-CoV-2 virus as well as Beta and Delta variants.
Time Frame: Study Days 1, 7, 28, 35 and 56
Population: Full Analysis Set: Includes all subjects from the Intent-to-Treat (ITT) set who received the prescribed study vaccine and underwent immunogenicity assessment at baseline and at least one time point after baseline.
Measure: Geometric Mean (95% Confidence Interval); unit: 50% neutralization titer
Arm/Group | Phase 1a, Group G1 | Phase 1a, Group G2 | Phase 1a, Group G3
Number analyzed (Participants) | 21 | 20 | 20
50% neutralization titer
  Ancestral, Day 1: number analyzed (Participants) | 21 | 19 | 20
  Ancestral, Day 1 | 6.0 [5.2 to 7.0] | 5.0 [4.2 to 5.9] | 5.0 [4.3 to 5.9]
  Ancestral, Day 7: number analyzed (Participants) | 21 | 19 | 20
  Ancestral, Day 7 | 6.7 [4.6 to 9.8] | 5.6 [3.8 to 8.4] | 5.0 [3.4 to 7.3]
  Ancestral, Day 28: number analyzed (Participants) | 19 | 18 | 18
  Ancestral, Day 28 | 13.3 [7.4 to 23.9] | 18.0 [9.9 to 32.9] | 5.0 [2.7 to 9.1]
  Ancestral, Day 35: number analyzed (Participants) | 17 | 17 | 16
  Ancestral, Day 35 | 12.6 [6.7 to 23.4] | 99.0 [53.2 to 184.2] | 5.0 [2.6 to 9.5]
  Ancestral, Day 56: number analyzed (Participants) | 14 | 16 | 12
  Ancestral, Day 56 | 5.4 [3.8 to 7.7] | 329.1 [236.9 to 457.2] | 5.0 [3.4 to 7.3]
  Beta, Day 1: number analyzed (Participants) | 21 | 19 | 20
  Beta, Day 1 | 5.4 [4.9 to 5.9] | 5.0 [4.6 to 5.5] | 5.0 [4.6 to 5.5]
  Beta, Day 28: number analyzed (Participants) | 19 | 18 | 17
  Beta, Day 28 | 8.8 [6.1 to 12.7] | 7.3 [5.0 to 10.6] | 5.2 [3.6 to 7.7]
  Beta, Day 35: number analyzed (Participants) | 16 | 17 | 16
  Beta, Day 35 | 7.8 [4.7 to 12.9] | 16.3 [10.0 to 26.5] | 5.0 [3.0 to 8.3]
  Beta, Day 56: number analyzed (Participants) | 14 | 16 | 12
  Beta, Day 56 | 5.0 [3.5 to 7.2] | 28.0 [20.0 to 39.2] | 5.0 [3.4 to 7.4]
  Delta, Day 1: number analyzed (Participants) | 21 | 19 | 20
  Delta, Day 1 | 5.4 [4.9 to 6.0] | 5.0 [4.5 to 5.6] | 5.0 [4.5 to 5.5]
  Delta, Day 28: number analyzed (Participants) | 18 | 18 | 18
  Delta, Day 28 | 10.8 [7.2 to 16.3] | 14.3 [9.5 to 21.6] | 5.0 [3.3 to 7.5]
  Delta, Day 35: number analyzed (Participants) | 17 | 17 | 16
  Delta, Day 35 | 9.7 [6.0 to 15.6] | 27.6 [17.2 to 44.5] | 5.0 [3.1 to 8.2]
  Delta, Day 56: number analyzed (Participants) | 14 | 16 | 12
  Delta, Day 56 | 5.7 [3.8 to 8.5] | 49.4 [33.8 to 72.0] | 5.0 [3.2 to 7.7]

5. Secondary Outcome: Geometric Mean Titer (GMT) of Spike Protein Binding Antibody in Serum (Phase 1a)
Description: Binding of serum antibody to SARS-CoV-2 spike protein was determined at baseline and post-vaccination by enzyme-linked immunosorbent assay (ELISA). Antibody levels are expressed as ELISA laboratory units (ELU)/mL. Binding antibody was tested against the spike protein of the ancestral (Wuhan) SARS-CoV-2 virus.
Time Frame: Study Days 1, 7, 28, 35, 56 and 112
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA laboratory units per mL
Arm/Group | Phase 1a, Group G1 | Phase 1a, Group G2 | Phase 1a, Group G3
Number analyzed (Participants) | 21 | 20 | 20
ELISA laboratory units per mL
  Day 1: number analyzed (Participants) | 20 | 19 | 20
  Day 1 | 28.4 [24.6 to 32.7] | 25.2 [21.7 to 29.1] | 25.2 [21.8 to 29.0]
  Day 7: number analyzed (Participants) | 20 | 19 | 20
  Day 7 | 33.4 [24.0 to 46.5] | 25.2 [18.0 to 35.3] | 25.2 [18.1 to 35.0]
  Day 28: number analyzed (Participants) | 17 | 18 | 18
  Day 28 | 161.5 [90.3 to 288.7] | 123.9 [70.5 to 217.9] | 25.2 [14.3 to 44.2]
  Day 35: number analyzed (Participants) | 15 | 17 | 16
  Day 35 | 186.8 [93.3 to 374.0] | 793.8 [413.5 to 1523.9] | 25.2 [12.8 to 49.3]
  Day 56: number analyzed (Participants) | 13 | 16 | 12
  Day 56 | 96.6 [65.6 to 142.3] | 4046.6 [2854.7 to 5736.2] | 25.2 [16.8 to 37.6]
  Day 112: number analyzed (Participants) | 1 | 3 | 3
  Day 112 | 127.0 [29.4 to 548.4] | 766.3 [329.3 to 1783.2] | 25.2 [10.8 to 58.5]

6. Secondary Outcome: Geometric Mean Titer (GMT) of Neutralizing Antibody in Serum (Phase 1b)
Description: as for outcome 4
Time Frame: Study Days 1, 7, 14, 28, 56, 84 and 168
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 50% neutralization titer
Arm/Group | Phase 1b, Group G4 | Phase 1b, Group G5
Number analyzed (Participants) | 27 | 26
50% neutralization titer
  Ancestral, Day 1 | 247.9 [163.7 to 375.4] | 196.3 [128.6 to 299.7]
  Ancestral, Day 7: number analyzed (Participants) | 26 | 26
  Ancestral, Day 7 | 353.5 [236.9 to 527.4] | 184.0 [123.4 to 274.6]
  Ancestral, Day 14 | 476.6 [336.8 to 674.4] | 209.9 [147.4 to 299.0]
  Ancestral, Day 28: number analyzed (Participants) | 27 | 25
  Ancestral, Day 28 | 404.3 [286.4 to 570.7] | 154.4 [107.9 to 220.9]
  Ancestral, Day 56: number analyzed (Participants) | 19 | 18
  Ancestral, Day 56 | 474.4 [263.5 to 854.0] | 194.5 [106.3 to 355.9]
  Ancestral, Day 84: number analyzed (Participants) | 6 | 4
  Ancestral, Day 84 | 323.7 [95.6 to 1095.5] | 264.2 [59.4 to 1175.8]
  Ancestral, Day 168: number analyzed (Participants) | 3 | 2
  Ancestral, Day 168 | 382.5 [177.0 to 826.5] | 429.8 [167.3 to 1104.2]
  Beta, Day 1 | 100.9 [66.4 to 153.4] | 62.2 [40.6 to 95.3]
  Beta, Day 7: number analyzed (Participants) | 26 | 25
  Beta, Day 7 | 215.1 [152.6 to 303.4] | 63.8 [44.9 to 90.5]
  Beta, Day 28: number analyzed (Participants) | 27 | 25
  Beta, Day 28 | 388.0 [263.0 to 572.5] | 63.9 [42.7 to 95.8]
  Beta, Day 56: number analyzed (Participants) | 19 | 18
  Beta, Day 56 | 267.9 [147.3 to 487.2] | 50.7 [27.4 to 93.6]
  Beta, Day 84: number analyzed (Participants) | 6 | 4
  Beta, Day 84 | 351.1 [118.6 to 1039.6] | 79.6 [21.1 to 300.6]
  Beta, Day 168: number analyzed (Participants) | 3 | 2
  Beta, Day 168 | 264.8 [147.2 to 476.2] | 139.6 [68.0 to 286.5]
  Delta, Day 1 | 65.0 [44.1 to 95.7] | 57.1 [38.5 to 84.6]
  Delta, Day 7: number analyzed (Participants) | 26 | 26
  Delta, Day 7 | 102.7 [70.7 to 149.3] | 54.3 [37.4 to 79.0]
  Delta, Day 28: number analyzed (Participants) | 27 | 25
  Delta, Day 28 | 138.5 [94.2 to 203.6] | 49.8 [33.4 to 74.4]
  Delta, Day 56: number analyzed (Participants) | 19 | 18
  Delta, Day 56 | 110.9 [65.9 to 186.6] | 39.6 [23.2 to 67.7]
  Delta, Day 84: number analyzed (Participants) | 6 | 4
  Delta, Day 84 | 221.2 [81.7 to 598.9] | 82.7 [24.4 to 280.3]
  Delta, Day 168: number analyzed (Participants) | 3 | 2
  Delta, Day 168 | 151.4 [59.0 to 388.8] | 201.9 [63.6 to 640.8]

7. Secondary Outcome: Geometric Mean Titer (GMT) of Spike Protein Binding Antibody in Serum (Phase 1b)
Description: as for outcome 5
Time Frame: Study Days 1, 7,14, 28, 56, 84,168 and 336
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA laboratory units per mL
Arm/Group | Phase 1b, Group G4 | Phase 1b, Group G5
Number analyzed (Participants) | 27 | 26
ELISA laboratory units per mL
  Day 1 | 5169.1 [3569.7 to 7485.0] | 3979.4 [2728.8 to 5803.1]
  Day 7: number analyzed (Participants) | 26 | 26
  Day 7 | 6952.7 [4915.7 to 9833.7] | 3894.4 [2753.4 to 5508.2]
  Day 14 | 8716.8 [6388.1 to 11894.3] | 3771.4 [2747.5 to 5176.8]
  Day 28: number analyzed (Participants) | 27 | 25
  Day 28 | 8915.0 [6489.2 to 12247.7] | 3269.2 [2350.2 to 4547.7]
  Day 56: number analyzed (Participants) | 19 | 18
  Day 56 | 8223.0 [5247.0 to 12820.8] | 3177.6 [2013.4 to 5105.0]
  Day 84: number analyzed (Participants) | 6 | 3
  Day 84 | 10090.9 [3840.3 to 26515.2] | 4718.2 [1445.2 to 15404.1]
  Day 168: number analyzed (Participants) | 3 | 2
  Day 168 | 8340.2 [4014.1 to 17328.5] | 6736.9 [2751.0 to 16497.5]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 1 year (Day 1 to Day 336) or early withdrawal, in all participants, in all groups.
Groups:
- Phase 1a, Group G1: Participants received VBI-2902a at a dose of 5 μg of S protein at Day 1 and placebo at Day 28
  VBI-2902a: VBI-2902a is an intramuscular injection of VBI-2902a investigational enveloped virus-like particle COVID-19 vaccine with aluminum phosphate adjuvant.
  Placebo: 0.9% sodium chloride
- Phase 1a, Group G2: Participants received VBI-2902a at a dose of 5 μg of S protein at Days 1 and 28
  VBI-2902a: VBI-2902a is an intramuscular injection of VBI-2902a investigational enveloped virus-like particle COVID-19 vaccine with aluminum phosphate adjuvant.
- Phase 1a, Group G3: Participants received placebo at Days 1 and 28
  Placebo: 0.9% sodium chloride
- Phase 1b, Group G4: Participants received VBI-2905a at a dose of 5 μg of S protein at Day 1
  VBI-2905a: VBI-2905a is an intramuscular injection of VBI-2905a investigational enveloped virus-like particle COVID-19 vaccine with aluminum phosphate adjuvant.
- Phase 1b, Group G5: Participants received placebo at Day 1
  Placebo: 0.9% sodium chloride
Arm/Group | Phase 1a, Group G1 | Phase 1a, Group G2 | Phase 1a, Group G3 | Phase 1b, Group G4 | Phase 1b, Group G5
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/20 | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/20 | 1/20 | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 16/21 | 17/20 | 15/20 | 27/27 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1a, Group G1 (N=21) | Phase 1a, Group G2 (N=20) | Phase 1a, Group G3 (N=20) | Phase 1b, Group G4 (N=27) | Phase 1b, Group G5 (N=26)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a, Group G1 (N=21) | Phase 1a, Group G2 (N=20) | Phase 1a, Group G3 (N=20) | Phase 1b, Group G4 (N=27) | Phase 1b, Group G5 (N=26)
Nausea (Gastrointestinal disorders) | 1 | 3 | 1 | 3 | 1
Chills (General disorders) | 2 | 3 | 2 | 1 | 1
Fatigue (General disorders) | 3 | 3 | 5 | 1 | 3
Injection site bruising (General disorders) | 1 | 2 | 0 | 0 | 0
Pain (General disorders) | 3 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 3 | 0 | 0
Vaccination site pain (General disorders) | 10 | 7 | 9 | 8 | 12
Vaccination site swelling (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 5 | 5 | 2 | 20 | 16
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Post vaccination syndrome (Injury, poisoning and procedural complications) | 3 | 5 | 6 | 3 | 4
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1 | 1
Headache (Nervous system disorders) | 3 | 5 | 4 | 2 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 4 | 5
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 1 | 2
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT04773665/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT04773665/SAP_001.pdf